CLINICAL TRIAL: NCT01538069
Title: Comparison Between Exercise Training and CPAP Treatment for Patients With Heart Failure and Sleep Apnea.
Brief Title: Heart Failure and Sleep Apnea: Exercise Training and Continuous Positive Airway Pressure
Acronym: CPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, Associate Professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP1226/11
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure; Sleep Apnea Syndromes
Keywords: Heart failure; Sleep apnea syndromes; Exercise; Continuous Positive Airway Pressure
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (No Intervention)
- Exercise group (Experimental)
  Interventions: Other: Exercise training
- CPAP group (Experimental)
  Interventions: Other: CPAP group
- Exercise and CPAP group (Experimental)
  Interventions: Other: Exercise and CPAP group

INTERVENTIONS:
Other: Exercise training — It consisted of three sessions/week, on non-consecutive days. The aerobic protocol consisted of a warm-up (strengthening exercises, 10 minutes), aerobic exercise (30 minutes in the first month and 45 minutes in the last two months) and cool-down (strengthening exercises, 10 minutes). The aerobic exercise intensity was established by heart rate levels that corresponded to anaerobic threshold, 10 heart rates down and 10 heart rates up, assessed by cardiopulmonary exercise testing. The strength training consisted of eight exercises attending the major muscle groups and the intensity was determined by 50-60% of one-repetition maximum (1-RM) and the progression of the training will be monthly: first month (a series of 12 repetitions with 50% 1-RM), second month (1 set of 15 repetitions with 60% 1-RM) and third months (2 sets of 10 repetitions with 60% 1-RM).
  Arms: Exercise group
Other: CPAP group — The CPAP treatment will be according to protocol of the Department of Psychobiology. Titration will be perform after randomization with ventilation device servo-assisted so as to ensure positive pressure within the first 24 hours of treatment. The treatment will be for three months.
  Arms: CPAP group
Other: Exercise and CPAP group — The patients randomized for this group will perform both Exercise protocol and CPAP treatment at the same time for three months.
  Arms: Exercise and CPAP group

SUMMARY:
Introduction. Heart failure is the result of primary ventricular dysfunction followed by neurohormorais changes, distribution of cardiac output, peripheral circulation, the skeletal and respiratory muscles, which determine their clinical and prognosis. Despite the advancement in treatment, morbidity and mortality remain high. Physical training appears as a therapeutic strategy, because most of its beneficial effects is by inducing changes in peripheral physiological changes resulting from heart failure. Associated factors that may contribute to its progression and worse prognosis, now beginning to be studied, such as sleep apnea, the diagnosis provides important prognostic information and a potential therapeutic option for these patients.

Objectives. Demonstrate the benefits of physical training for patients with heart failure and sleep apnea, and compare treatment with CPAP alone and associated with the exercise program. Will also be assessed risk and adherence to physical training.

Material and Methods. The design will be prospective, longitudinal, randomized consecutive patients. After screening and baseline evaluations the patients will be randomized into Group 1 (CPAP, n = 20), Group 2 (CPAP + Physical training, n = 20), Group 3 (Physical Training, n = 20) and Group 4 (Control without intervention, n = 20). Outcomes (baseline and 3 months): Quality of sleep (polysomnography), Quality of life (Minnesota and SF-36), sexual function (QS-M and QS-F) and functional capacity (cardiopulmonary exercise testing and isokinetic testing). Physical training: aerobic and resistance exercises three times a week for three months. CPAP therapy:after polysomnography for titration with ventilator servo-assisted, and outpatient follow monthly, for three months.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-70 years
* New York Heart Association Class II-III
* Clinically stable for one month
* Ejection fraction <40%
* Peak VO2 <20 ml/kg/min
* Stable and optimized medical therapy at least one month before the study
* B-blocker therapy
* Clinical and polysomnographic diagnosis of sleep apnea (IAH>10)

Exclusion Criteria:

* Patients with previous treatment of sleep apnea
* New York Heart Association Class IV
* Clinical instability
* Poor adherence to drug treatment
* Myocardial infarction or revascularization within the past two months
* Unstable angina
* Symptomatic arrhythmias (pacemaker and defibrillator)
* Obstructive aortic or mitral valvular disease
* Hypertrophic cardiomyopathy
* Abnormal exercise testing
* Pulmonary arterial pressure >50mmHg
* Chronic obstructive pulmonary disease
* Intermittent leg claudication
* Musculoskeletal disorders or psychiatric disease that prevents the patient from understanding and following the exercise prescription safely

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Polysomnography | Two evaluations (baseline and 3 month)
  To evaluate changes from Baseline in quality of sleep, mainly sleep apnea, after 3 months. Overnight polysomnography will be perform using a digital system with 17 channels(EMBLA, Medicare Medical Devices). The following variables will be monitor: electroencephalogram, electrooculogram, electromyogram, electrocardiogram,snoring and body position. Airflow will be monitor using a thermocouple and pressure transducer. Chest and abdominal piezo-sensors will monitor respiratory effort. Arterial oxygen saturation and pulse will be record with a pulse oxymeter.

SECONDARY OUTCOMES:
Cardiopulmonary exercise testing | Two evaluations (baseline and 3 month)
  To evaluate changes from Baseline in functional capacity, after 3 months. All patients will realize a symptom limited, treadmill test with respiratory gas exchange analysis, according to Weber protocol. Heart rate and rhythm were monitored by 12-lead electrocardiogram. Blood pressure was determined by a mercury sphygmomanometer at rest and at the end of each stage. The self-perceived level of exertion (15-point Borg scale) was assessed at peak effort.
Isokinetic strength and endurance | Two evaluations (baseline and 3 month)
  To evaluate changes from Baseline in strenght and endurance of legs after 3 months. Strength and endurance of the knee extensors and flexors were measured using an isokinetic dynamometer, which modifies the speed and angle of movements. The test protocol consisted of a warm-up (five minutes on a cycle ergometer), three repetitions at 60degree/second (Maximal dynamic strength, peak torque - Nm) and 10 repetitions at 180degree/second (endurance, total work - J), followed by a cool-down (five minutes on a cycle ergometer).
Quality of Life | Two evaluations (baseline and 3 month)
  To evaluate changes from Baseline in quality of life after 3 months. Quality of life will be measure by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) that assesses disease-specific health-related quality of life by including the patient's perception of the effects of chronic heart failure and its treatment on daily life. And by 36-item Short-Form Health Survey (SF-36) that is a generic instrument to evaluate the quality of life.
Sexual Function | Two evaluations (baseline and 3 month)
  To evaluate changes from Baseline in sexual function after 3 months. Sexual function of men will be evaluate by the questionnaire Quociente Sexual Masculino (QS-M) and sexual function of women will be evaluate by the questionnaire Quociente Sexual Feminino (QS-F). Both questionnaires evaluate the sexual function of men and women in a comprehensive way to measure the elements of physical, emotional and relational.

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Servantes, PT, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Bittencourt L, Javaheri S, Servantes DM, Kravchychyn ACP, Almeida DR, Tufik S. In patients with heart failure, enhanced ventilatory response to exercise is associated with severe obstructive sleep apnea. J Clin Sleep Med. 2021 Sep 1;17(9):1875-1880. doi: 10.5664/jcsm.9396. PMID 33949944